CLINICAL TRIAL: NCT00033306
Title: A Phase II Study Of Epothilone Analog BMS-247550 In Patients With Metastatic Colorectal Cancer Previously Treated With A Fluoropyrimidine And Irinotecan
Brief Title: BMS-247550 in Treating Patients With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069272; UAB-0145; BMS-CA163-012; UAB-F011029021; NCI-G02-2051
Record Dates: First submitted 2002-04-09; First posted 2003-08-06 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — ixabepilone; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BMS-247550 (Experimental)
  Interventions: Drug: ixabepilone; Drug: Fluoropyrimidine; Drug: Irinotecan

INTERVENTIONS:
Drug: ixabepilone
Drug: Fluoropyrimidine
Drug: Irinotecan

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of BMS-247550 in treating patients who have metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical activity of BMS-247550, as measured by the tumor response rate, in patients with metastatic colorectal cancer previously treated with a fluoropyrimidine and irinotecan.
* Determine the safety of this drug in these patients.
* Determine the response duration, time to progression, and survival in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive BMS-247550 IV over 1 hour on days 1-5. Treatment repeats every 21 days for up to 18 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive up to 4 additional courses of treatment beyond CR.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 19-55 patients will be accrued for this study within 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic colorectal adenocarcinoma
* Prior treatment for metastatic disease with at least:

  * One regimen of irinotecan in combination with a fluoropyrimidine OR
  * Two regimens comprising fluoropyrimidine-based first-line therapy and irinotecan-based second-line therapy

    * May have received cetuximab and/or a fluoropyrimidine as part of second- line therapy
* Disease progression during or within 4 months of treatment with irinotecan
* At least 1 bidimensionally measurable lesion
* No known CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 2,000/mm^3
* Platelet count greater than 125,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT no greater than 2.5 times ULN (5 times ULN if hepatic metastases present)

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No New York Heart Association class III or IV heart disease
* No history of unstable angina, myocardial infarction, or congestive heart failure within the past 6 months

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known prior severe hypersensitivity reactions to agents containing Cremophor EL
* No motor or sensory neuropathy grade 2 or greater
* No concurrent serious uncontrolled infection or other nonmalignant medical illness
* No concurrent psychiatric disorders or other conditions that would preclude study compliance
* No other active malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No concurrent immunotherapy
* No growth factors for 24 hours before and after cytotoxic chemotherapy

Chemotherapy:

* See Disease Characteristics
* Additional prior adjuvant or neoadjuvant chemotherapy allowed
* At least 4 weeks since prior chemotherapy and recovered
* No more than 2 prior regimens of cytotoxic chemotherapy for metastatic disease
* No prior oxaliplatin
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy except hormone replacement therapy

Radiotherapy:

* At least 3 weeks since prior radiotherapy and recovered
* No prior radiotherapy to target lesion unless the lesion has shown progression after completion of radiotherapy
* No concurrent therapeutic radiotherapy

  * Focal radiotherapy for palliation of bone symptoms may be allowed

Surgery:

* At least 1 week since prior minor surgery (3 weeks for major surgery) and recovered

Other:

* No other concurrent experimental anticancer medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2002-02; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Determine the clinical activity of BMS-247550, as measured by the tumor response rate, in patients with metastatic colorectal cancer previously treated with a fluoropyrimidine and irinotecan. | baseline to survival

SECONDARY OUTCOMES:
Determine the safety of this drug in these patients. | baseline to survival
Determine the response duration, time to progression, and survival in patients treated with this drug. | baseline to survival

CONTACTS AND LOCATIONS:
Overall Officials: Andres Forero-Torres, MD, CSU, Study Chair — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Georgia Cancer Specialists, Atlanta, Georgia